CLINICAL TRIAL: NCT03483688
Title: A Phase Ⅰb Study Evaluating Safety and Efficacy of Anti-CD19 Chimeric Antigen Receptor T-cell (C-CAR011) Treatment in Subjects With Relapsed or Refractory B-Cell Non-Hodgkin Lymphoma
Brief Title: A PhaseⅠb Study Evaluating Safety and Efficacy of C-CAR011 Treatment in B- NHL Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Shanghai AbelZeta Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBMG-C2017007
Record Dates: First submitted 2018-03-14; First posted 2018-03-30 (Actual); Last update posted 2020-03-05 (Actual); Status verified 2018-03

CONDITIONS: B-cell Non-Hodgkin Lymphoma
Keywords: B-cell Non-Hodgkin Lymphoma; Refractory; Relapsed
MeSH Terms: conditions — Lymphoma, B-Cell; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD19-directed CAR-T cells (Experimental): Lymphocytes will be transduced with lentiviral vector containing CAR-CD19 gene
  Interventions: Biological: CD19-directed CAR-T cells

INTERVENTIONS:
Biological: CD19-directed CAR-T cells — CD19-directed CAR-T cells single infusion intravenously at a target dose of 0.5-5.0 x 10^6 anti-CD19 CAR+ T cells/kg
  Other Names: Anti-CD19 chimeric antigen receptor T cells (C- CAR011)

SUMMARY:
This is a single arm, single-center, non-randomized study to evaluate the safety and efficacy of C-CAR011 therapy in relapsed or refractory B cell Non-Hodgkin Lymphoma (NHL).

DETAILED DESCRIPTION:
The study will include the following sequential phases: Screening, Pre- Treatment (Cell Product Preparation; Lymphodepleting Chemotherapy), Treatment and Follow-up

ELIGIBILITY:
Inclusion Criteria:

* Volunteered to participate in this study and signed informed consent.
* Age 18-70 years old, male or female.
* Relapse or refractory B cell non-Hodgkin's lymphoma ,Histologically diagnosed as DLBCL,follicular lymphoma and Mantle cell lymphoma according to the NCCN. nonHodgkin's lymphoma Clinical Practice Guidelines (2017 Version 1)

  1. DLBCL and Follicular Lymphoma (stage Ⅲ-Ⅳ, grade Ⅲb).

     1. Progressive disease after the last standard chemotherapy regimens.
     2. Stable disease after the last standard chemotherapy regimens(at least 4 cycles of first-line therapy or 2 cycles of later-line therapy).
     3. Relapse or progressive disease within 12 months after autologous stem cell transplantation (SCT).
  2. Follicular lymphoma (stage Ⅲ-Ⅳ) (gradeⅠ-Ⅲa)

     1. Relapse or progressive disease within 1 year after the last standard chemotherapy regimens(At least 2 combination chemotherapy regimens).
     2. Stable disease after the last standard chemotherapy regimens(at least 2 cycles of combination chemotherapy regimens).
  3. Mantle cell lymphoma

     1. Relapse after 1st CR or persistent disease, and not eligible or appropriate for SCT.
     2. Relapse or progressive disease within 1 year after the last chemotherapy regimens(at least 4 cycles of first-line therapy or 2 cycles of later- line therapy).
     3. Relapse or progressive disease within 12 months after autologous SCT.
* All subjects must have received anti-CD20 monoclonal antibody (unless tumor is CD20-negative) and anthracycline-containing chemotherapy regimens according to NCCN non-Hodgkin lymphoma Clinical Practice Guidelines (2017 Version 1).
* At least one measurable lesion per revised IWG Response Criteria (the longest diameter of the tumor ≥ 1.5cm).
* Expected survival ≥ 12 weeks.
* ECOG score 0-1.
* Left ventricular ejection fraction (LVEF) ≥ 50% (detected by echocardiography).
* No active pulmonary infections, normal pulmonary function and oxygen saturation ≥ 92% on room air.
* At least 2 weeks from receiving previous treatment (radiotherapy or chemotherapy) prior to leukapheresis.
* No contraindications of leukapheresis.
* Female subjects in childbearing age, their serum or urine pregnancy test must be negative, and must agree to take effective contraceptive measures during the trial.

Exclusion Criteria:

* History of allergy to cellular products.
* Laboratory tests: absolute neutrophil count < 1.0 × 10^9 /L, platelet count < 50×10^9 /L, serum albumin < 30 g/L,serum bilirubin > 1.5 ULN, serum creatinine > ULN, ALT/AST > 3 ULN.
* History of CAR T cell therapy or any other genetically modified T cell therapy.
* Relapse after allogeneic hematopoietic stem cell transplantation.
* Active infections that require treatment (uncomplicated urinary tract infections and bacterial pharyngitis are allowed), prophylactic antibiotic, antiviral and antifungal treatment are permitted.
* Hepatitis B or hepatitis C virus infection (including carriers), syphilis, as well as acquired or congenital immune deficiency diseases, including but not limited to HIV infection.
* Class III or IV heart failure according to the NYHA Heart Failure Classifications.
* QT interval prolongation ≥ 450 ms.
* History of epilepsy or other central nervous system disorders.
* Evidence of CNS lymphoma by head enhancement scan or magnetic resonance imaging.
* History of other primary cancers, with the following exceptions.

  1. Excisional non-melanoma (e.g. cutaneous basal cell carcinoma).
  2. Cured in situ carcinoma (e.g. cervical cancer, bladder cancer, breast cancer).
* Autoimmune diseases that require treatment, immune deficiency diseases or other diseases that require immunosuppressive therapy.
* Used of systemic steroids within two weeks (using inhaled steroids is an exception).
* Women who are pregnant or lactating, or who have breeding intent in 6 months.
* Participated in any other clinical trial within three months.
* Any situation that investigators believe the risk of the subjects is increased or results of the trial are disturbed.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-03-06 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
AE | 12 weeks
  Incidence of adverse events (AEs) and serious adverse events (SAEs)

SECONDARY OUTCOMES:
Overall response rate (ORR) | 12 months
  The ORR will be assessed at weeks 4 ，weeks 12 ，months 6 and months 12
Duration of remission (DOR) | 12 months
  The DOR will be assessed at months 12
Progression free survival (PFS) | 12 months
  The PFS will be assessed at months 12
Overall survival rate（OSR） | 12 months
  The OSR will be assessed at weeks 12 ，months 6 and months 12

CONTACTS AND LOCATIONS:
Overall Officials: Daobin Zhou, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Zhang L, Zhang Y, Zhou DB. [Anti-CD19 CART (C-CAR011) Therapy for Relapsed or Refractory B-Cell Non-Hodgkin Lymphoma]. Zhongguo Shi Yan Xue Ye Xue Za Zhi. 2021 Aug;29(4):1141-1147. doi: 10.19746/j.cnki.issn.1009-2137.2021.04.019. Chinese. PMID 34362494